CLINICAL TRIAL: NCT05068609
Title: Nivolumab in the Real World in Patients With Squamous Cell Carcinoma of the Head & Neck (SCCHN) - Patient Reported Outcomes (PRO)
Brief Title: A Study of Nivolumab in Participants With Squamous Cell Carcinoma of the Head & Neck (SCCHN) - Patient Reported Outcomes (PRO)
Acronym: VOLUME-PRO
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-7F9
Record Dates: First submitted 2021-09-08; First posted 2021-10-06 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: BMS-936558; Health Related Quality of Life; Metastatic; Nivolumab; Opdivo®; Patient Reported Outcomes; Recurrent; Squamous Cell Carcinoma of the Head and Neck; VOLUME-PRO
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Neoplasm Metastasis; Recurrence | interventions — Nivolumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort 1: Participants with squamous cell carcinoma of the head and neck (SCCHN) treated with nivolumab
  Interventions: Biological: Nivolumab

INTERVENTIONS:
Biological: Nivolumab — Participants in this study are being treated with nivolumab for SCCHN
  Other Names: Opdivo®, BMS-936558

SUMMARY:
The purpose of the study is to capture the utilization of nivolumab among participants with squamous cell carcinoma of the head and neck (SCCHN) since its approval, and to describe the health related quality of life (HRQoL) among participants treated with nivolumab in a real-world setting.

DETAILED DESCRIPTION:
This is a phase 4 prospective chart review study with patient reported outcome (PRO) administration. The study population consists of participants diagnosed with squamous cell carcinoma of the head and neck (SCCHN) and are being treated with nivolumab. Eligible participants will be enrolled and observed from enrollment up to eight weeks. Demographic and clinical characteristics will be collected at enrollment. PROs will be administered at enrollment and again at a follow-up standard of care visit approximately eight weeks after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of recurrent/metastatic squamous cell carcinoma of the head and neck (SCCHN)
* Age ≥18 years at time of nivolumab treatment initiation
* Investigator has decided that nivolumab is appropriate therapy and the participant had received at least one administration of nivolumab for the treatment of recurrent/metastatic SCCHN prior to enrolment in the study
* Charts/records include treatment start date of nivolumab
* Provide consent and is willing to self-complete on-site patient reported outcomes (PROs) on at least one occasion

Exclusion Criteria:

* Currently enrolled in an interventional clinical trial for their SCCHN
* Received systemic treatment for any other primary cancer within 6 months of study enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population for this study will be approximately 50 adult participants, with a diagnosis of recurrent or metastatic squamous cell carcinoma of the head and neck (SCCHN) currently being treated with nivolumab in the United Kingdom, Switzerland, Spain, or Canada. The study population will include participants with available data from medical records at enrollment who are willing to complete patient reported outcome (PRO) assessments.
Sampling Method: Non-Probability Sample
Enrollment: 509 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2021-10-18 (Actual); Study Completion 2021-10-18 (Actual)

PRIMARY OUTCOMES:
Distribution of demographic characteristics of R/M SCCHN participants treated with nivolumab: Month and year of birth | At enrollment
  Recurrent/Metastatic (R/M) Squamous Cell Carcinoma of the Head & Neck (SCCHN)
Distribution of demographic characteristics of R/M SCCHN participants treated with nivolumab: Sex | At enrollment
Distribution of demographic characteristics of R/M SCCHN participants treated with nivolumab: Race/ethnicity | At enrollment
Distribution of demographic characteristics of R/M SCCHN participants treated with nivolumab: Smoking status | At enrollment
Distribution of clinical characteristics of R/M SCCHN participants treated with nivolumab: Primary tumor location | At enrollment
Distribution of clinical characteristics of R/M SCCHN participants treated with nivolumab: Metastasis locations | At enrollment
Distribution of clinical characteristics of R/M SCCHN participants treated with nivolumab: Histology | At enrollment
Distribution of clinical characteristics of R/M SCCHN participants treated with nivolumab: Date of diagnosis of R/M SCCHN | At enrollment
Distribution of clinical characteristics of R/M SCCHN participants treated with nivolumab: Stage at locally advanced/metastatic SCCHN diagnosis | At enrollment
Distribution of patterns of use of nivolumab treatment in participants with R/M SCCHN: Duration of nivolumab therapy | Up to 8 weeks following enrollment
Distribution of patterns of use of nivolumab treatment in participants with R/M SCCHN: Drug discontinuation | Up to 8 weeks following enrollment
Distribution of doses of nivolumab therapy in participants with R/M SCCHN | Up to 8 weeks following enrollment
Distribution of subsequent treatment in participants discontinuing nivolumab | Up to 8 weeks following enrollment
Distribution of patient reported health-related quality of life (HRQoL) measures through European Organisation for Research and Treatment of Cancer Quality of Life- Core Questionnaire in participants treated with nivolumab for R/M SCCHN | At enrollment, Up to 8 weeks
Distribution of patient reported HRQoL measures through EQ-5D-5L in participants treated with nivolumab for R/M SCCHN | At enrollment, Up to 8 weeks
Distribution of patient reported HRQoL measures through European Organisation for Research and Treatment of Cancer Head and Neck Cancer Module in participants treated with nivolumab for R/M SCCHN | At enrollment, Up to 8 weeks
Distribution of patient reported HRQoL measures through CTSQ in participants treated with nivolumab for R/M SCCHN | At enrollment, Up to 8 weeks
  Cancer Therapy Satisfaction Questionnaire (CTSQ)
Distribution of patient reported HRQoL measures through WPAI:GH in participants treated with nivolumab for R/M SCCHN | At enrollment, Up to 8 weeks
  Work Productivity and Activity Impairment Questionnaire: General Health (WPAI:GH)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Mount Laurel, New Jersey, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome